CLINICAL TRIAL: NCT05521178
Title: A Multicenter, Prospective Cohort Study for Detection of Cardiotoxicities in Patients Receiving Ibrutinib or Acalabrutinib for CLL
Brief Title: Cardiotoxicities in Patients Receiving BTKi
Status: Withdrawn | Type: Observational
Why Stopped: Funding for study was withdrawn
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Inhye Ahn, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 22-301
Record Dates: First submitted 2022-08-28; First posted 2022-08-30 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Electrocardiography; Echocardiography; Blood Pressure Monitoring, Ambulatory; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples With DNA: Samples retained, with potential for extraction of DNA from at least one of the types of samples retained (e.g., frozen tissue, whole blood)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ibrutinib: Patients receiving ibrutinib for the treatment of CLL.
  Interventions: Diagnostic Test: Electrocardiogram; Diagnostic Test: Echocardiogram; Diagnostic Test: Cardiac magnetic resonance imaging; Device: Mobile cardiac telemetry; Diagnostic Test: Blood pressure monitoring; Diagnostic Test: Blood draw
- Acalabrutinib: Patients receiving acalabrutinib for the treatment of CLL.
  Interventions: Diagnostic Test: Electrocardiogram; Diagnostic Test: Echocardiogram; Diagnostic Test: Cardiac magnetic resonance imaging; Device: Mobile cardiac telemetry; Diagnostic Test: Blood pressure monitoring; Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Electrocardiogram — ECG to monitor electrical activities of the heart on each visit
  Other Names: ECG
Diagnostic Test: Echocardiogram — Echocardiogram at baseline and 6 months
  Other Names: TTE
Diagnostic Test: Cardiac magnetic resonance imaging — Cardiac MRI at baseline and 6 months
  Other Names: Cardiac MRI
Device: Mobile cardiac telemetry — Mobile cardiac telemetry at baseline and 6 months
  Other Names: Mobile telemetry
Diagnostic Test: Blood pressure monitoring — Home blood pressure monitoring three times per week
  Other Names: Home blood pressure monitoring
Diagnostic Test: Blood draw — Blood draw at baseline, 3 and 6 months

SUMMARY:
This is a multicenter, prospective, observational cohort study to comprehensively and longitudinally evaluate and characterizes the cardiovascular events with CLL patients who are initiating treatment with a Bruton's tyrosine kinase (BTK) inhibitor ibrutinib or acalabrutinib.

DETAILED DESCRIPTION:
This research study includes three visits for research blood, physical exam, and cardiac testing at baseline, 3 months, and 6 months. The study will collect the following data during the 6-month study period:

* Blood sample collection
* Electrocardiogram (ECG)
* Echocardiogram
* Cardiac magnetic resonance imaging (MRI)
* Mobile cardiac telemetry
* Blood pressure measurement

ELIGIBILITY:
Inclusion criteria

* Patients with confirmed diagnosis of CLL who are planned to start either ibrutinib or acalabrutinib per standard of care, in monotherapy or in combination with an anti-CD20 antibody, venetoclax, and/or a PI3K inhibitor. Both treatment-naïve and relapsed or refractory CLL are allowed.
* No known history of paroxysmal, persistent, or permanent atrial fibrillation. Exception: The study allows enrollment of up to 10 patients with a known history of paroxysmal atrial fibrillation (exploratory cohort).
* No known history chronic symptomatic congestive heart failure or documented ejection fraction < 50%.
* Creatinine ≤ 1.5x institutional upper limit of normal (ULN). An adequate kidney function is necessary to ensure safety of IV contrast given before cardiac MRI.
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%).

Exclusion criteria

* Prior exposure to ibrutinib or acalabrutinib.
* Patients with a clinical contraindication to MRI.
* Patients with childbearing potential who cannot or do not wish to use an effective method of contraception, during the study period and for 12 months after the final treatment used for the purposes of the study.
* Patients with any medical condition, psychiatric condition, or social situation that in the opinion of the investigator would compromise compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed diagnosis of CLL who are planned to start either ibrutinib or acalabrutinib per standard of care, in monotherapy or in combination with an anti-CD20 antibody, venetoclax, and/or a PI3K inhibitor. Both treatment-naïve and relapsed or refractory CLL are allowed.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of atrial arrhythmias | During 6 months of BTK inhibitor therapy
  Any documented evidence of atrial arrhythmia including symptomatic and asymptomatic events captured by EKG, 28-day mini cardiac telemetry, or monitoring of cardiac rhythm during echocardiogram or cardiac MRI.

SECONDARY OUTCOMES:
Incidence of ventricular arrhythmias | During 6 months of BTK inhibitor therapy
  Assessed by 28-day mobile telemetry
Severity of ventricular arrythmia | During 6 months of BTK inhibitor therapy
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Inhye Ahn, MD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu